CLINICAL TRIAL: NCT02228928
Title: Efficacy and Safety of 0.625% and 1.25% Capsaicin Patch in the Management of Peripheral Neuropathic Pain ; Early Phase II, Multi-center, Randomized, and Semi-double Blind Controlled Clinical Trial
Brief Title: Study of Capsaicin Patch for the Management of Peripheral Neuropathic Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Samyang Biopharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAPNP201
Record Dates: First submitted 2014-08-26; First posted 2014-08-29 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2014-09

CONDITIONS: Peripheral Nerve Injury; Postherpetic Neuralgia
Keywords: Peripheral Nerve Injury; Postherpetic Neuralgia
MeSH Terms: conditions — Peripheral Nerve Injuries; Neuralgia, Postherpetic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- CAPNP, 50 ug/cm2 capsaicin patch (Experimental): 50 ug/cm2 capsaicin patch, 49cm2, 1patch/4days
  Interventions: Drug: CAPNP, 50 ug/cm2 capsaicin patch
- CAPNP, 100 ug/cm2 capsaicin patch (Experimental): 100ug/cm2 capsaicin patch, 49cm2, 1patch/4days
  Interventions: Drug: CAPNP, 100 ug/cm2 capsaicin patch
- 0.075% capsaicin cream (Active Comparator): capsaicin cream qc/day
  Interventions: Drug: 0.075% capsaicin cream
- Placebo patch (Placebo Comparator)
  Interventions: Other: Placebo patch

INTERVENTIONS:
Drug: CAPNP, 50 ug/cm2 capsaicin patch
  Arms: CAPNP, 50 ug/cm2 capsaicin patch
Drug: CAPNP, 100 ug/cm2 capsaicin patch
  Arms: CAPNP, 100 ug/cm2 capsaicin patch
Drug: 0.075% capsaicin cream
  Arms: 0.075% capsaicin cream
Other: Placebo patch
  Arms: Placebo patch

SUMMARY:
The efficacy and safety of the low concentration [0.65% (50 µg/cm2) and 1.25% (100 µg/cm2)] capsaicin patches and compared them to conventional 0.075% capsaicin cream and placebo patch in patients suffering from peripheral neuropathy

ELIGIBILITY:
Inclusion Criteria:

* patients who are 18 years of age or older aged having chronic peripheral neuropathy related with a diagnosis of either PHN or DPN
* patients with chronic peripheral neuropathic pain for more than 3 months with an 11-pointed Numeric Rating Scale (NRS) pain score ≥ 4
* patients with a diagnosis of PHN were eligible if at least 3 months had elapsed since shingles vesicle crusting
* patients with DPN and well controlled diabetes were asked to maintain a stable dose of oral hypoglycemic or insulin during the study period
* patients taking concomitant pain medications such as anticonvulsants, antidepressants, anxiolytics, and opioids including tramadol were required to maintain a stable dose for at least 4 weeks before the study enrollment
* any conservative therapies such as TENS, physical therapy, chiropractic, massage, biofeedback, or yoga were stopped at least 5 weeks before the enrollment
* women of childbearing age were required to have a negative pregnancy test and were to be willing to use an effective method of contraception for at least 28 days after the last exposure to study medication

Exclusion Criteria:

* diffusely distributed neuropathic pain resulting from spinal stenosis, postoperative origin, complex regional pain syndrome, or genetic neurological disease, or significant pain outside the target area
* significant pain of an etiology other than PHN or DNP
* other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or with investigational product administration or may interfere with compliance or the interpretation of study results andin the judgment of the investigator would make the subject inappropriate to participate in the study
* painful PHN areas located on the face or above the scalp hairline
* an implanted medical device for the treatment of neuropathic pain
* use of topically applied agents including capsaicin-containing products, a 5% lidocaine patch or similar products, local anesthetics, or steroids within the past 21 days
* hypersensitivity known to capsaicin; current use of any class 1 anti-arrhythmic drug; and uncontrolled diabetes mellitus or uncontrolled hypertension
* If patients have taken oral NSAID or COX2 Inhibitor, it should be stopped at least2 weeks before randomization; however acetaminophen for pain control was allowed up to 4g per day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Mean difference in the change of daily NRS pain score | 6 weeks
  Mean numeric change in numerical rating scale pain score from the baseline (Visit 2) to the score at weeks 6 (Visit 5) in each group

SECONDARY OUTCOMES:
Percentage of patients with >=30% or >=50% reduction in pain | 6 weeks
  The percentage of responders (>=30% reduction) and the percentage of patients achieving a >=50% in NRS pain scores were compared among groups
Daily Sleep Interference Scale | 2, 4, 6 weeks
Clinical Global Impression for Improvement | 2, 4, 6 weeks
  Clinical Global Impression of Change by the physician and Patient Global Impression of Change by the patients were used to evaluate the subjective perception of decrease in pain intensity
EQ-5D | 6 weeks
  For EQ-5DTM Health Survey, mean change from the baseline (Visit 2) to the score at weeks 6 (Visit 5) was shown as frequencies and their percentages

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoula National University Bundang Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Moon JY, Lee PB, Kim YC, Lee SC, Nahm FS, Choi E. Efficacy and Safety of 0.625% and 1.25% Capsaicin Patch in Peripheral Neuropathic Pain: Multi-Center, Randomized, and Semi-Double Blind Controlled Study. Pain Physician. 2017 Feb;20(2):27-35. PMID 28158151